CLINICAL TRIAL: NCT02184182
Title: Liver Resection After Portal Vein Ligation / Embolization and Transection Plane Devascularization With Radio Frequency / Microwave: Pilot Study on Primary and Secondary Liver Tumors
Brief Title: Laparoscopic Microwave Ablation and Portal Vein Ligation for Staged Hepatectomy (LAPS)
Acronym: LAPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, full professor of general surgery, MD, PhD, Azienda Ospedaliera di Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2934P
Record Dates: First submitted 2014-06-23; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Liver Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VLS ablation/portal ligation/hepatectomy (Experimental): Step1:
  * exploratory laparoscopy to exclude extrahepatic disease
  * right portal vein ligation if surgically feasible
  * RF/MW ablation on the future line of transection (of segment 4 close to left lateral lobe)
  * radiological portal embolization within 48h form the laparoscopic procedure if the right portal vein ligation is not feasible CT volumetric scan to evaluate the left lateral lobe hypertrophy after 9±2 from Step 1
  Step 2: only if FRL/body weight > 0.5
  - laparoscopic/laparotomic right trisectionectomy
  Interventions: Procedure: VLS ablation/portal ligation/hepatectomy

INTERVENTIONS:
Procedure: VLS ablation/portal ligation/hepatectomy — Step1:
  * exploratory laparoscopy to exclude extrahepatic disease
  * right portal vein ligation if surgically feasible
  * RF/MW ablation on the future line of transection (of segment 4 close to left lateral lobe)
  * radiological portal embolization within 48h form the laparoscopic procedure if the right portal vein ligation is not feasible
  CT volumetric scan to evaluate the left lateral lobe hypertrophy after 9±2 from Step 1
  Step 2: only if FRL/body weight > 0.5
  - laparoscopic/laparotomic right trisectionectomy
  Other Names: VLS Ablation & Portal Vein Ligation for Staged Hepatectomy

SUMMARY:
One of the limiting factors in the execution of a liver resection, in particular an extended liver resection, it's represented by the future remnant liver (FRL) after hepatic surgery. In cases of normal organ function an FRL of 25% is considered sufficient. In case of impaired hepatic function or a history of chemotherapy, it is considered safe if at least of 40%.

Many strategies have been developed and proposed to increase the resectability in patients undergoing major liver resections.

One of these is a new two-stage technique proposed recently by a group of German surgeons. This approach consists in the ligation of the right portal vein associated with resection of the liver along the falciform ligament (step 1). Step 2, after a period of 9 days (median - 5-25 days), after a volumetric CT to ensure an adeguate hypertrophy of the left lateral lobe due to the combination of right portal occlusion and segment 4 devascularization, the patient undergo a right trisectionectomy. The hypertrophy of the left lateral lobe is shown to be of 74%, higher than any other techniques of ligation or portal embolizatiol proposed in the literature.

On the basis of the clinical experiences reported the investigators designed a new protocol of two-stage hepatic resection for the treatment of primary or secondary tumors of the right lobe. Step1: laparoscopic radio frequency / microwave ablation of the future transection plane between segment 4 and left lateral lobe and surgical ligation or embolization of the right portal vein. The ablation has the purpose to devascularize the segment 4 and has the same significance of the resection of the liver along the falciform ligament described by the Regensburg group.

Step2: After a period of time of 9 ± 2 days, following a volumetric CT showing an adequate liver volume gain (ratio FRL / patient body weight> 0.5), the patient undergo the second-stage surgery: laparoscopic/ laparotomic right trisectionectomy.

DETAILED DESCRIPTION:
In patients with primary or metastatic liver tumors, the only potentially curative therapeutic option is represented by hepatic resection. Nowdays extended resections can be performed with acceptable morbidity and mortality. There is no unanimous definition on the criteria of resectability and the ability to perform a more or less extensive liver resection is deferred to the expertise of the center and the surgical team. The investigators will consider a tumor resectable if the surgical procedure does not damage vital structures, the normal function of the organ is preserved and and the tumor is completely removed (R0 resection). One of the limiting factors in the execution of a liver resection, in particular if it is extended, it's represented by the future remnant liver (FRL) after hepatic resection. In cases of normal organ function an FRL of 25% is considered sufficient. In case of impaired hepatic function or a history of chemotherapy, it is considered safe if at least of 40%.

Many methods have been developed and proposed to increase the resectability in patients undergoing major liver resections. In case of bilobar tumor, a two-step approach (two-stage hepatectomy)have been proposed. This procedure implies that one of the two lobes is initially freed of disease by tumor resection or ablation. After achieving an adequate compensatory hypertrophy of the lobe freed by the tumor (usually 4-6 weeks),a contralateral liver resection can be done to treat the remnant tumor.

To increase the FRL another approach is to occlude the portal branches towards one of liver lobes. This can be done with a surgical ligation (laparotomy or laparoscopy) or radiologically, using portal embolization. The technique allows to increase from 10% to 46% of the FRL with the possibility of obtaining a resection R-0 in 70-100% of cases. It is unclear whether there is any difference between the methods of portal occlusion (ligation vs embolization). To further increase hypertrophy after portal occlusion in liver tumors occupying the right liver, some researchers proposed to embolize the portal branches of segment 4th together with the right portal vein.

The group of Regensburg has introduced a new technique in two stages for tumors of the right lobe, which combines the methods mentioned above. This two-stage approach consists in the ligation of the right portal vein associated with resection of the liver along the falciform ligament (step 1). Step 2, after a period of 9 days (median - 5-25 days), after a volumetric CT to ensure an adeguate hypertrophy of the left lateral lobe, the patient undergo a right trisectionectomy. The hypertrophy of the left lateral lobe is shown to be of 74%, higher than any other techniques of ligation or portal embolizatiol proposed in the literature.

The rationale of this technique is the complete portal devascularization of the right lobe plus segment 4 that produce a greater stimulus to hypertrophy of the left lateral segments. This occurs in less time than other methods above described and allows to reduce the timeframe between the two steps and minimizes the risk of interprocedural progression of the underlying disease (incidence of drop outs in the two-stage hepatectomy of 20% for progression disease).

The morbidity of this two-stage approach was 44% (complications of Clavien grade III and IV) that mimics the data reported in the literature for extended hepatic resections (20-50%). The 12%mortality rate was similar to one described by Lang et al for left trisegmentectomies.

On the basis of the clinical experiences reported the investigators designed a new protocol of two-stage hepatic resection for the treatment of primary or secondary tumors of the right lobe. Step1: laparoscopic radio frequency / microwave ablation of the future transection plane between segment 4 and left lateral lobe and surgical ligation or embolization of the right portal vein. The ablation has the purpose to devascularize the segment 4 and has the same significance of the resection of the liver along the falciform ligament described by the Regensburg group.

Step2: After a period of time of 9 ± 2 days, following a volumetric CT showing an adequate liver volume gain (ratio FRL / patient body weight> 0.5), the patient undergo the second-stage surgery: laparoscopic/ laparotomic right trisectionectomy

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years (M and F)
* Liver tumors that interests the right hepatic lobe (segments 4,5,6,7,8) with possible involvement of the caudate lobe (segment 1) or bilobar disease with less than 3 lesions in the left lateral lobe without vascular involvement and amenable to surgically resectable or ablation in the Step1.
* Absence of extrahepatic disease
* Normal hepatic function (total bilirubin <3 mg / dL)
* Performance status: ECOG 0
* In case of liver cirrhosis MELD score <9
* Patients without prior chemotherapy or with previous chemotherapy but with response disease
* Patients who give their consent to the intervention

Exclusion Criteria:

* CT Evidence of involvement of the major vessels in the future remnant liver
* Presence of more than 3 nodules in the left lateral lobe
* Presence of extrahepatic disease
* Severe hepatic impairment
* Age> 70 years
* Previous liver surgery (prior liver resections)
* Patient receiving chemotherapy with documented disease progression

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of R0 resections | 30days after Step2
  Percentage of operations in which a complete oncological radicality (R0) is achived

SECONDARY OUTCOMES:
Perioperative mortality (3 months) | 3 moths
  Percentage of perioperative mortality (3 months)
Perioperative complication (Clavien Classification) | 1 month
  Percentage of perioperative complication described using Clavien Dindo Classification
Time to progression | 12 months
Overall survival | 12 and 24 months
  Overall survival at 12 and 24 months after surgery
disease free survival | 12 months
hepatic diesease free survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Cillo, MD PhD, Study Chair — Azienda Ospedaliera di Padova
Locations (1):
- Chirurgia Epatobiliare e Trapianto Epatico - Azienda Ospedaliera di Padova, Padua, Padova, Italy

REFERENCES:
- [Background] Schnitzbauer AA, Lang SA, Goessmann H, Nadalin S, Baumgart J, Farkas SA, Fichtner-Feigl S, Lorf T, Goralcyk A, Horbelt R, Kroemer A, Loss M, Rummele P, Scherer MN, Padberg W, Konigsrainer A, Lang H, Obed A, Schlitt HJ. Right portal vein ligation combined with in situ splitting induces rapid left lateral liver lobe hypertrophy enabling 2-staged extended right hepatic resection in small-for-size settings. Ann Surg. 2012 Mar;255(3):405-14. doi: 10.1097/SLA.0b013e31824856f5. PMID 22330038
- [Background] Lang H, Sotiropoulos GC, Brokalaki EI, Radtke A, Frilling A, Molmenti EP, Malago M, Broelsch CE. Left hepatic trisectionectomy for hepatobiliary malignancies. J Am Coll Surg. 2006 Sep;203(3):311-21. doi: 10.1016/j.jamcollsurg.2006.05.290. Epub 2006 Jul 13. PMID 16931303
- [Background] Jaeck D, Oussoultzoglou E, Rosso E, Greget M, Weber JC, Bachellier P. A two-stage hepatectomy procedure combined with portal vein embolization to achieve curative resection for initially unresectable multiple and bilobar colorectal liver metastases. Ann Surg. 2004 Dec;240(6):1037-49; discussion 1049-51. doi: 10.1097/01.sla.0000145965.86383.89. PMID 15570209
- [Background] Farges O, Belghiti J, Kianmanesh R, Regimbeau JM, Santoro R, Vilgrain V, Denys A, Sauvanet A. Portal vein embolization before right hepatectomy: prospective clinical trial. Ann Surg. 2003 Feb;237(2):208-17. doi: 10.1097/01.SLA.0000048447.16651.7B. PMID 12560779
- [Background] Tartter PI. The association of perioperative blood transfusion with colorectal cancer recurrence. Ann Surg. 1992 Dec;216(6):633-8. doi: 10.1097/00000658-199212000-00004. PMID 1466616
- [Background] Donati M, Stavrou GA, Oldhafer KJ. Current position of ALPPS in the surgical landscape of CRLM treatment proposals. World J Gastroenterol. 2013 Oct 21;19(39):6548-54. doi: 10.3748/wjg.v19.i39.6548. PMID 24151380
- [Background] Lang H, Sotiropoulos GC, Fruhauf NR, Domland M, Paul A, Kind EM, Malago M, Broelsch CE. Extended hepatectomy for intrahepatic cholangiocellular carcinoma (ICC): when is it worthwhile? Single center experience with 27 resections in 50 patients over a 5-year period. Ann Surg. 2005 Jan;241(1):134-43. doi: 10.1097/01.sla.0000149426.08580.a1. PMID 15622001
- [Background] Are C, Iacovitti S, Prete F, Crafa FM. Feasibility of laparoscopic portal vein ligation prior to major hepatectomy. HPB (Oxford). 2008;10(4):229-33. doi: 10.1080/13651820802175261. PMID 18806869
- [Background] de Santibanes E, Alvarez FA, Ardiles V. How to avoid postoperative liver failure: a novel method. World J Surg. 2012 Jan;36(1):125-8. doi: 10.1007/s00268-011-1331-0. PMID 22045448
- [Background] van Lienden KP, Hoekstra LT, Bennink RJ, van Gulik TM. Intrahepatic left to right portoportal venous collateral vascular formation in patients undergoing right portal vein ligation. Cardiovasc Intervent Radiol. 2013 Dec;36(6):1572-1579. doi: 10.1007/s00270-013-0591-5. Epub 2013 Mar 13. PMID 23483283
- See also: Online resource of Chirurgia Epatobiliare e Trapianto Epatico, Università degli Studi di Padova — http://www.fegatochirurgia.com